CLINICAL TRIAL: NCT06620289
Title: The Impact of Dental Desensitization Visits Facilitated by a Child Life Specialist on Pediatric Patients' Distress and Cooperation
Brief Title: Impact of Dental Desensitization Facilitated by a Child Life Specialist Distress and Cooperation
Status: Enrolling by invitation | Type: Observational
Sponsor: Children's Hospital Colorado (Other)
Responsible Party: Principal Investigator, Stephanie Barta, Senior Certified Child Life Specialist, Children's Hospital Colorado
Other Study IDs: 24-0196
Record Dates: First submitted 2024-09-25; First posted 2024-10-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Desensitization; Dental Anxiety; Dental Care; Distress, Emotional; Cooperation, Patient
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Dental Desensitization Clinic — The goal of offering desensitization visits is to reduce the dental anxiety and distress of patients and enhance their cooperation during future appointments. The specifics of the desensitization are individualized to meet the unique needs of each patient based on information provided by the parent/caregiver. A standard desensitization visit involves providing the patient the opportunity to sit in the exam chair; touch the toothbrush and rubber prophy cup, mouth mirror, fluoride applicator brush, air-water syringe tip and saliva ejector tip; gain exposure to the dental lights and sounds commonly experienced in the dental visit; practice opening their mouth; and tolerate toothbrush and rubber prophy cup, mirror, explorer, fluoride applicator brush, air-water syringe, and salvia ejector in the mouth. If the child is unable or unwilling to participate, these activities are modeled on the parent or by the CCLS.

SUMMARY:
The aim of this study is to evaluate whether dental desensitization visits facilitated by a Certified Child Life Specialist (CCLS) significantly impact pediatric patients' distress and cooperation levels from the start of desensitization visit(s) to end of the desensitization visit(s), end of desensitization visit to start of subsequent hygiene appointment, and end of hygiene appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patients and parents of patients aged 2-25 years who have been referred to the desensitization clinic.
* Patients who meet with a CCLS for dental desensitization.

Exclusion Criteria:

* Patients younger than 2 years old and older than 25 years old.

Ages: 2 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric patients and their parents scheduled in the dental center at Children's Hospital Colorado Health Pavillion referred to a child life specialist-facilitated desensitization clinic will be recruited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Frankl Behavioral Rating Scale (FBRS) | From enrollment to the end of study at approximately 3 months.
  The FBRS is widely used in pediatric dentistry to evaluate patient behavior. FBRS consists of four behavior categories ranging from "definitely positive" to "definitely negative," with higher scores indicating more cooperation. The rating is assigned by the treating pediatric provider and recorded in the patient's medical record at the end of the visit. Participants achieve a scored on a scale ranging from 1 (definitely negative) to 4 (definitely positive).

SECONDARY OUTCOMES:
Pre-Visit Parent Survey | Before desensitization visit.
  Parents/caregivers will be asked to fill out a questionnaire before and after the desensitization visit and after the subsequent hygiene appointment. Questions will relate to previous dental experience, previous visit Sensory Tolerance Checklist and the parent's perception of visit success.
Repeated Desensitization Visit - Pre-Desensitization Parent Survey | Before repeated (if applicable) desensitization visits.
  If a patient requires more than one dental desensitization visit during the study period, the research team will collect data during subsequent desensitization visits. This survey is a modified and shortened version of the "Pre-Visit Parent Survey" and aims to assess if there have been any changes to the child's developmental diagnoses as well as track how many desensitization visits the patient has had.
Sensory Tolerance Checklist | From enrollment to the end of study at approximately 3 months.
  Tolerance is operationalized as allowing dental instrument(s) to touch a patient for 1-2 seconds without resisting or exhibiting distress. Three attempts will be made for each step on the checklist before being identified as incomplete. This checklist will be completed by the CCLS and the clinical research coordinator (CRC) for interrater reliability during the desensitization visit.
The Children's Fear Scale (CFS) | From enrollment to the end of study at approximately 3 months.
  Measure fear in children undergoing painful medical procedures. Patients receive a score ranging from 0 (Not scared at all) to 5 (Most scared possible).
Psychosocial Risk Assessment in Pediatrics (PRAP) | From enrollment to the end of study at approximately 3 months.
  The PRAP assesses pediatric patients by evaluating which patients are at risk of experiencing elevated distress during their health care encounters. Children are scored on a cumulative risk score from 0 (low risk) to 24 (high risk). Scores are categorized into low (0-7 points), medium (8-14 points), and high (15-24) risk levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No